CLINICAL TRIAL: NCT06527105
Title: The Effects of Non-pharmacological Interventions on the Quality of Sleep in Cardiac Surgical Patients
Brief Title: Impact of Sleep Quality on Outcomes After Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amrita Institute of Medical Sciences & Research Center (Other)
Responsible Party: Principal Investigator, Nagarjuna P, Assistant Professor, Department of Cardiac Anesthesia, Amrita Institute of Medical Sciences & Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IEC-AIMS-2023-CARDANES-009
Record Dates: First submitted 2024-07-23; First posted 2024-07-30 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Sleep; Atrial Fibrillation; Delirium, Postoperative; Complications, Postoperative
Keywords: Cardiac surgery; Sleep quality
MeSH Terms: conditions — Atrial Fibrillation; Emergence Delirium; Postoperative Complications; Sleep Initiation and Maintenance Disorders | interventions — Ear Protective Devices

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Active Comparator): Eye masks and Ear plugs given during sleep
  Interventions: Device: Eye masks and ear plugs
- Control group (No Intervention): Routine care given without any intervention

INTERVENTIONS:
Device: Eye masks and ear plugs — Eye masks and ear plugs given during sleeping time in Icu After cardiac surgery
  Arms: Interventional group

SUMMARY:
Sleep is a basic human need and is essential for good quality of life, good health. In fact, humans spend one third of their life time in sleeping or attempting to do so. However, sleep is not given due importance in intensive care unit (ICU)'s, although it is critical in healing process. Patient's usually get admitted to the hospital few days prior to the surgery, for complete evaluation, depending on the procedure planned. Hospital environment being, an entirely new place for inpatients, will invariably affect their sleep. Sleep deprivation is one of the major sources of anxiety and stress in all the patients during ICU stay. This means that most of patients are sleep deprived, by the time they are admitted to ICU.

The negative effects of sleep deprivation include postoperative brain dysfunction like inattention, restlessness, hallucinations, agitation, aggressiveness. The degree of cognitive impairment may range from subtle derangements in attention, reason, clarity of thought and capacity of decision making to confusion and delirium. Sleep deprivation can also induce hypertension, fatigue, metabolic disorders, cerebrovascular and cardiovascular disease

ELIGIBILITY:
Inclusion Criteria:

* Adult cardiac surgical patients aged above 18years undergoing elective cardiac surgery

Exclusion Criteria:

* Not willing to give consent
* Preoperative sleep medications use
* Preoperative psychological disorders, on mechanical ventilation for >12hrs, dementia, cerebrovascular accident

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Quality of sleep | 6 months
  On the morning after the intervention, patient's sleep quality will be assessed using Richard-Campbell sleep questionnaire (RCSQ). Each point in RCSQ will be scored using a visual analog score, ranging from 0-100. Total score will be calculated and then will be divided by 5.

SECONDARY OUTCOMES:
Atrial fibrillation | 6 months
  Postoperative atrial fibrillation
Delirium | 6 months
  Postoperative Delirium
Intensive care unit stay | 6 months
  Duration of intensive care unit stay (in hours to days)
Vasoactive inotropic score | 6 months
  Vasoactive inotropic score is calculated by multiplying the dose of each vasoactive drug used with 10. (minimum score is 0, while maximum score can go upto 20. Higher the score worse is the outcome
Mechanical ventilation | 6 months
  Duration of mechanical ventilation (hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Nagarjuna, Kochi, Kerala, India

IPD SHARING:
Plan to Share IPD: No